CLINICAL TRIAL: NCT07082699
Title: The Efficacy of Antegrade and Retrograde Enemas in the Management of Low Anterior Resection Syndrome and Improving the Rate of Ileostomy Reversal: A Single-Centre, Prospective Randomised Controlled Trial
Brief Title: The Efficacy of Antegrade and Retrograde Enemas Management in Low Anterior Resection Syndrome and Improving the Rate of Ileostomy Reversal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Hui Yang, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT2024153
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: LARS - Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard of care (No Intervention)
- antegrade enema (Experimental)
  Interventions: Other: antegrade enema
- retrograde enema (Experimental)
  Interventions: Other: retrograde enema

INTERVENTIONS:
Other: antegrade enema — Introduce saline at a flow rate of 40 ml/minute through the distal end of the ileostomy. The initial enema volume is approximately 500 ml, with a maximum of 1000 ml. Perform twice weekly for one month.
  Arms: antegrade enema
Other: retrograde enema — Introduce saline at a flow rate of 40 ml/minute through the anus. The initial enema volume is approximately 500 ml, with a maximum of 1000 ml. Perform twice weekly for one month.
  Arms: retrograde enema

SUMMARY:
Anterior rectal resection has become the primary surgical treatment for rectal cancer. However, studies have reported that up to 80%-90% of patients who undergo anterior rectal resection experience varying degrees of defecation dysfunction after surgery, such as frequent bowel movements, urgent bowel movements, and faecal incontinence, known as low anterior resection syndrome (LARS). This can lead to a decline in quality of life after surgery and even partial loss of social functioning.

ELIGIBILITY:
Inclusion Criteria:

1. According to the NCCN guidelines for the pathological diagnosis of rectal cancer, the patient has primary rectal adenocarcinoma;
2. Age ≥ 18 years;
3. Previously underwent rectal resection with prophylactic ileostomy via laparoscopy, robotics, or open surgery;
4. Expected to undergo ileostomy reversal surgery within 1-2 months;
5. Possesses normal cognitive and communication abilities;
6. Voluntarily participates in this study and has signed an informed consent form.

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) classification III or higher;
2. Concurrent inflammatory bowel disease, Crohn's disease, or other intestinal diseases;
3. Mental disorders, long-term use of psychiatric drugs;
4. Contraindications to enemas.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of ileostomy reversal | Two months after the last enema
low anterior resection syndrome score (LARS score) | Evaluations were conducted one day before enema, one month after enema, one month, two months, three months, and six months after stoma closure.
  The LARS score consists of five components and the total score, ranging from 0 to 42. Severity levels are categorized as follows: no LARS (0-20 points), minor LARS (21-29 points), and major LARS (30-42 points).

SECONDARY OUTCOMES:
quality of sleep | Evaluations were conducted one day before enema, one month after enema, one month, two months, three months, and six months after stoma closure.
  Quality of sleep was evaluated by Pittsburgh Quality Index (PSQI). The PSQI assesses a participant's sleep quality in the previous month using 18 items divided into 7 components. Each component is graded between 0 and 3. The total score is 0-21, with higher scores indicating poorer sleep quality.
bowel function | one month, two months, three months, and six months after stoma closure.
  The Memorial Sloan-Kettering Cancer Center Bowel Function Instrument (MSKCC BFI) is used to assess bowel function. This questionnaire comprises three dimensions, totaling 18 items. The total scale score ranged from 18 to 90, with higher scores indicating better bowel function.
cancer patients' quality of life | one month, two months, three months, and six months after stoma closure.
  The quality of life was assessd by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29). The scale includes 4 functional domains, 19 symptom domains, and 6 stoma-related items. Each item, except for item 18 (which indicates the presence or absence of a stoma), is rated on a 4-point scale: 'not at all,' 'a little,' 'quite a bit,' and 'very much,' corresponding to scores of 1 to 4, respectively. Scores are converted into standardized values ranging from 0 to 100 using polarization. Higher scores in the functional domains indicate better function, whereas higher scores in the symptom domains reflect more severe symptoms.

OTHER OUTCOMES:
The psychosocial adjustment level of patients with enterostomy | Evaluate one day before starting enemas and one month after enemas before performing stoma closure.
  The psychosocial adjustment level of patients with enterostomy were evaluated using the Ostomy Adjustment Inventory-20 (OAI-20). OAI-20 adopts a 5-level Likert scoring method, forward scores range from 0 (strongly disagree) to 4 (strongly agree), while reverse scores range from 4 (strongly disagree) to 0(strongly agree). Total scores range from 0 to 80, where scores <40 indicate low psychosocial adjustment, scores between 40 and 59 indicate medium psychosocial adjustment, and scores ≥60 indicate high psychosocial adjustment levels.
The Stoma-Specific Quality of Life | Evaluate one day before starting enemas and one month after enemas before performing stoma closure.
  The Stoma-Specific Quality of Life-Questionnaire (Stoma QoL) was designed specifically for patients with ostomy and consists of 20 entries, each of which is divided into 4 levels: always, sometimes, rarely, never, with a score ranging from 1 to 4. The ratings range from 20 to 80, with higher levels indicating higher HRQoL.
Observation chart for anal excretion and irritation symptoms during ostomy (self-made) | Evaluate one day before starting enemas and one month after enemas before performing stoma closure
  This was designed to assess anal feces and discomfort sensations in stoma patients during their stoma time. The questionnaire consisted of four main questions dealing with frequency of defecation, perception of bowel movement, sensation of irritation in the anal region, and the patient's reaction to irritants. These four specific questions as follow:
  1. In the last week, how often have you felt discharge oozing from around your anus?
  2. In the last week, how often have you felt a bowel movement around your anus?
  3. In the last week, how often have you felt irritation in your bowel movements?
  4. Do you experience skin irritation or discomfort from anal discharge? (five-point scale: "very", "rather", "generally", "somewhat", "not at all")